CLINICAL TRIAL: NCT01532830
Title: Non-Invasive Neurostimulation of the Vagus Nerve With the GammaCore Device For the Relief of Symptoms Associated With Migraine
Brief Title: Non-Invasive Neurostimulation For the Relief of Symptoms Associated With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-US-01
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Migraine
Keywords: vagus nerve stimulation; vagal nerve stimulation; nVNS; VNS; migraine; non invasive; gammacore
MeSH Terms: conditions — Migraine Disorders

ARMS (1):
- Active (Experimental): n-VNS active therapy
  Interventions: Device: n-VNS

INTERVENTIONS:
Device: n-VNS
  Other Names: gammaCore

SUMMARY:
The purpose of this pilot study is to assess feasibility and clarify the design of future study(ies) to support marketing approval of the GammaCore™ device for the treatment and/or prevention of migraine symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 18 and 55 years.
* Has been previously diagnosed as suffering from migraine, in accordance with the ICHD-2 Classification criteria (2nd), with or without aura.
* Experiences at least 2 migraines per month, but less than 15 headache days per month (over the last 3 months).
* Has age of onset of migraine less than 50 years old.
* Is able to give written Informed Consent

Exclusion Criteria:

* Has a history of aneurysm, intracranial hemorrhage, brain tumors or significant head trauma.
* Has a lesion (including lymphadenopathy) at the GammaCore™ treatment site.
* Has known or suspected severe atherosclerotic cardiovascular disease, severe carotid artery disease (e.g. bruits or history of TIA or CVA), congestive heart failure (CHF), coronary artery disease or recent myocardial infarction.
* Has a history or baseline ECG that identifies the presence of a clinically significant unstable cardiac arrhythmia, second degree heart block type II, history of ventricular tachycardia or ventricular fibrillation, or known cardiac syndromes that may be associated with increased risk of sudden death in otherwise healthy people.
* Has had a previous bilateral or right cervical vagotomy.
* Has a clinically significant irregular heart rate or rhythm.
* Has uncontrolled high blood pressure.
* Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant.
* Has a history of carotid endarterectomy or vascular neck surgery on the right side.
* Has been implanted with metal cervical spine hardware or has a metallic implant near the GammaCore™ stimulation site.
* Has a recent or repeated history of syncope.
* Has a recent or repeated history of seizure.
* Has a history or suspicion of narcotic abuse.
* Takes medication for acute headaches more than 10 days per month.
* Is pregnant, nursing, thinking of becoming pregnant in the next 3 months, or of childbearing years and is unwilling to use an accepted form of birth control.
* Is participating in any other therapeutic clinical investigation or has participated in a clinical trial in the preceding 30 days.
* Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with follow-up requirements, or provide self-assessments is compromised (e.g., homeless, developmentally disabled, prisoner).
* Is a relative of or an employee of the investigator or the clinical study site.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UCSF Headache Center, San Francisco, California
  - New York Headache Center, New York, New York
  - Montefiore Headache Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goadsby PJ, Grosberg BM, Mauskop A, Cady R, Simmons KA. Effect of noninvasive vagus nerve stimulation on acute migraine: an open-label pilot study. Cephalalgia. 2014 Oct;34(12):986-93. doi: 10.1177/0333102414524494. Epub 2014 Mar 7. PMID 24607501

RESULTS

PARTICIPANT FLOW:
Groups:
- gammaCore Device: non-invasive vagus nerve stimulator gammaCore: treatment with gammaCore vagus nerve stimulator
Period: Overall Study
Arm/Group | gammaCore Device
Started | 30
Completed | 26
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: Randomized population
Arm/Group | Active
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 38.5 [19 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19
  Black | 3
  Hispanic | 6
  Asian | 1
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Safety - Number of Participants With Adverse Effects
Description: The primary outcome measure for this study was the assessment of adverse events as unanticipated or anticipated.
Time Frame: End of Study - 7 weeks
Population: Randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | Active
Number analyzed (Participants) | 30
Participants
  Unanticipated Adverse Effects | 0
  Anticipated Adverse Effects | 13

2. Secondary Outcome: Mean Change in Headache Pain From Baseline to 120 Minutes
Description: Headache was measured on a 4 point scale where 0 = no pain, 1 = mild, 2 = moderate, 3 = severe pain at baseline (start of attack), 5, 15, 30, 45, 60, 90 and 120 minutes.
  Data presented shows the average change from baseline to 120 minutes
Time Frame: 120 minutes
Population: Randomized population. 2 subjects were excluded from the analysis due to protocol deviations
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Active
Number analyzed (Participants) | 28
units on a scale
  Mean baseline pain score | 1.84 [0 to 3]
  Mean 120 minutes pain score | 1.20 [0 to 3]

3. Secondary Outcome: Change in Photophobia (Visual) From Baseline to 120 Minutes
Description: Presence of photophobia (yes or no) was captured at baseline and 120 minutes.
Time Frame: Base line and 120 minutes
Population: Randomized population. Data was missing for 3 patients
Measure: Number; unit: migraines with photophobia
Arm/Group | Active
Number analyzed (Participants) | 27
migraines with photophobia
  Migraine attacks with photophobia at baseline | 53
  Migraine attacks with photophobia at 120 minutes | 37

4. Secondary Outcome: Change in Phonophobia (Auditory) From Baseline to 120 Minutes
Description: Presence of phonophobia (yes or no) was captured at baseline and 120 minutes.
Time Frame: Baseline and 120 minutes
Population: Randomized population. Data was missing for 3 patients
Measure: Number; unit: migraines with phonophobia
Arm/Group | Active
Number analyzed (Participants) | 27
migraines with phonophobia
  Migraine attacks with phonophobia at baseline | 32
  Migraine attacks with phonophobia at 120 minutes | 15

5. Secondary Outcome: Mean Change in Nausea From Baseline to 120 Minutes
Description: Nausea was captured in the diary and measured on a 4 point scale, where 0 = no nausea, 1 = mild, 2 = moderate and 3 = severe nausea, at baseline and 120 minutes.
Time Frame: Baseline 120 minutes
Population: Randomized population. Data was missing for 3 patients
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Active
Number analyzed (Participants) | 27
units on a scale
  Nausea severity at baseline | 0.42 [0 to 3]
  Nausea severity at 120 minutes | 0.34 [0 to 3]

6. Secondary Outcome: Mean Change in Functional Disability
Description: Functional disability was captured in the diary and measured on a 4 point scale, where 0 = no disability, able to function normally and where 3 = performance of daily activities severely impaired, measured at baseline and 120 minutes.
Time Frame: Baseline and 120 minutes
Population: Randomized population. Data was missing for 3 patients
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Active
Number analyzed (Participants) | 27
units on a scale
  Mean disability score at baseline | 1.07 [0 to 3]
  Mean disability score at 120 minutes | 0.77 [0 to 3]

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | Active
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 13/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=30)
Stiff Neck (Musculoskeletal and connective tissue disorders) | 2 (4)
Viral Infection (Infections and infestations) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Discomfort to the neck into the upper right shoulder with tingling (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 2 (2)
Neck twitched a little during use of the device (Nervous system disorders) | 1 (1)
Lip drooping during use of the device (Nervous system disorders) | 1 (1)
Facial drooping (Nervous system disorders) | 1 (1)
Frequent urination (Renal and urinary disorders) | 1 (4)
Raspiness of voice (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neck redness (Skin and subcutaneous tissue disorders) | 1 (2)
Neck swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right shoulder spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tinnitus left ear (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less